CLINICAL TRIAL: NCT03088540
Title: A Global, Randomised, Phase 3, Open-label Study of REGN2810 (ANTI-PD 1 Antibody) Versus Platinum Based Chemotherapy in First Line Treatment of Patients With Advanced or Metastatic PD L1+Non-small Cell Lung Cancer
Brief Title: Study of REGN 2810 Compared to Platinum-Based Chemotherapies in Participants With Metastatic Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1624; 2016-004407-31 (EudraCT Number); 2024-511454-45-00 (Registry Identifier: EUCT Number)
Record Dates: First submitted 2017-03-03; First posted 2017-03-23 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma，Non-Small-Cell Lung; Lung Carcinomas, Non-Small-Cell; Non-small-cell Lung Carcinoma; Nonsmall Cell Lung Cancer
Keywords: Previous Smoker; Current Smoker; Stage IIIB; Stage IIIC; Stage IV; PD-L1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Paclitaxel; Gemcitabine; Cisplatin; Carboplatin; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard-of-care chemotherapy (Active Comparator): Standard-of-care chemotherapy will administered from these options:
  Doses of Paclitaxel + cisplatin OR Doses Paclitaxel + carboplatin OR Doses Gemcitabine + cisplatin or Doses Gemcitabine + carboplatin OR Doses Pemetrexed + cisplatin followed by optional pemetrexed maintenance OR Doses Pemetrexed + carboplatin followed by optional pemetrexed maintenance
  Interventions: Drug: Pemetrexed; Drug: Paclitaxel; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin
- cemiplimab (Experimental): cemiplimab regimen as monotherapy as per study protocol
  Interventions: Drug: cemiplimab

INTERVENTIONS:
Drug: Pemetrexed — Patients will be administered pemetrexed chemotherapy as per protocol with either cisplatin or carboplatin
  Arms: Standard-of-care chemotherapy
Drug: Paclitaxel — Patients will be administered paclitaxel chemotherapy as per protocol with either cisplatin or carboplatin
  Arms: Standard-of-care chemotherapy
Drug: Gemcitabine — Patients will be administered gemcitabine chemotherapy as per protocol with either cisplatin or carboplatin
  Arms: Standard-of-care chemotherapy
Drug: Cisplatin — Administered with either Pemetrexed, Paclitaxel or gemcitabine.
  Arms: Standard-of-care chemotherapy
Drug: Carboplatin — Administered with either Pemetrexed, Paclitaxel or gemcitabine.
  Arms: Standard-of-care chemotherapy
Drug: cemiplimab — Patients will be administered cemiplimab as per protocol.
  Other Names: REGN2810; Libtayo
  Arms: cemiplimab

SUMMARY:
The primary objectives of the study are:

* To compare the overall survival (OS) of cemiplimab versus standard-of-care platinum-based chemotherapies in the first-line treatment of patients with advanced or metastatic non-small cell lung cancer (NSCLC) whose tumors express PD-L1 in ≥50% of tumor cells
* To compare the progression-free survival (PFS) of cemiplimab versus standard-of-care platinum-based chemotherapies in the first-line treatment of patients with advanced or metastatic NSCLC whose tumors express PD-L1 in ≥50% of tumor cells

The key secondary objective of the study is to compare the objective response rate (ORR) of cemiplimab versus platinum-based chemotherapies

DETAILED DESCRIPTION:
There is option to join genomics sub-study.

ELIGIBILITY:
Key Inclusion Criteria:

A patient must meet the following criteria to be eligible for inclusion in the study:

1. Patients with histologically or cytologically documented squamous or non squamous NSCLC with stage IIIB or stage IIIC disease who are not candidates for treatment with definitive concurrent chemoradiation or patients with stage IV disease who received no prior systemic treatment for recurrent or metastatic NSCLC
2. Archival or newly obtained formalin-fixed tumor tissue from a metastatic/recurrent site, which has not previously been irradiated
3. Tumor cells expressing PD L1 above a specific percentage of tumor cells by IHC performed by the central laboratory
4. At least 1 radiographically measureable lesion per RECIST 1.1
5. ECOG performance status of ≤1
6. Anticipated life expectancy of at least 3 months
7. Adequate organ and bone marrow function

Key Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

1. Patients that have never smoked, defined as smoking <100 cigarettes in a lifetime
2. Active or untreated brain metastases or spinal cord compression
3. Patients with tumors tested positive for EGFR gene mutations, ALK gene translocations, or ROS1 fusions
4. Encephalitis, meningitis, or uncontrolled seizures in the year prior to randomization
5. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management. A history of radiation pneumonitis in the radiation field is permitted as long as pneumonitis resolved ≥6 months prior to randomization
6. Patients with active, known, or suspected autoimmune disease that has required systemic therapy in the past 2 years
7. Patients with a condition requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 14 days of randomization
8. Another malignancy that is progressing or requires treatment
9. Uncontrolled infection with hepatitis B or hepatitis C or human immunodeficiency virus (HIV) or diagnosis of immunodeficiency
10. Active infection requiring systemic therapy within 14 days prior to randomization
11. Prior therapy with anti-PD 1 or anti-PD L1
12. Treatment-related immune-mediated AEs from immune-modulatory agents
13. Receipt of an investigational drug or device within 30 days
14. Receipt of a live vaccine within 30 days of planned start of study medication
15. Major surgery or significant traumatic injury within 4 weeks prior to first dose
16. Documented allergic or acute hypersensitivity reaction attributed to antibody treatments
17. Known psychiatric or substance abuse disorder that would interfere with participation with the requirements of the study, including current use of any illicit drugs
18. Pregnant or breastfeeding women
19. Women of childbearing potential or men who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 6 months after the last dose

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death, assessed up to 68 months
Progression-free survival (PFS) as assessed by a blinded Independent review committee (IRC) using RECIST 1.1 | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 68 months
  PFS as assessed by a blinded IRC using RECIST 1.1.

SECONDARY OUTCOMES:
Objective response rates (ORR) | From date of randomization to the date of the first objectively documented progression or the date of subsequent anti-cancer therapy, whichever comes first, up to 68 months
  The number of patients with a best overall response (BOR) of confirmed Complete Response (CR) or Partial Response (PR) divided by the number of patients in the efficacy analysis set
Best overall response (BOR) | From date of randomization until the date of first documented progression or the date of subsequent anti-cancer therapy, whichever came first, assessed up to 68 months
  The BOR, as determined by the IRC per RECIST 1.1
Compare the duration of response (DOR) of cemiplimab versus platinum based chemotherapies | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 68 months
  Duration of response will be defined as the time between the date of first response (CR or PR) to the date of the first documented tumor progression (per RECIST 1.1) or the date of subsequent anti-cancer therapy or death due to any cause, whichever comes first
Change from baseline in quality of life (QoL) scores as assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Baseline up to 26 months after treatment
Change from baseline in in lung cancer symptom scores as measured by the EORTC Lung Cancer 13 (EORTC QLQ-LC13) | Baseline up to 26 months after treatment
Incidence of Adverse Events (AEs) | Baseline up to 68 months after treatment
Incidence of serious adverse events (SAEs) | Baseline up to 68 months after treatment
Incidence of deaths | Baseline up to 68 months after treatment
Incidence of laboratory abnormalities | Baseline up to 68 months after treatment
  Number of patients with laboratory abnormalities
Measure concentrations of cemiplimab in serum | Baseline up to 68 months after treatment
  Maximum Plasma Concentration [Cmax]
Characterize the pharmacokinetics (PK) of cemiplimab | Baseline up to 68 months after treatment
  Area Under the Curve [AUC]

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (192):
- Australia (3):
  - Clinical Study Site, Albury, New South Wales
  - Clinical Study Site, Wollongong, New South Wales
  - Clinical Study Site, Fitzroy
- Belarus (2):
  - Clinical Study Site, Minsk
  - Clinical Study Site, Mogilev
- Brazil (19):
  - Clinical Study Site 1, Porto Alegre, Rio Grande do Sul
  - Clinical Study Site, Barretos
  - Clinical Study Site, Curitiba
  - Clinical Study Site, Joinville
  - Clinical Study Site, Lajeado
  - Clinical Study Site, Mogi das Cruzes
  - Clinical Study Site, Passo Fundo
  - Clinical Study Site, Pelotas
  - Clinical Study Site 2, Porto Alegre
  - Clinical Study Site 3, Porto Alegre
  - Clinical Study Site, Recife
  - Clinical Study Site, Rio de Janeiro
  - Clinical Study Site, Salvador
  - Clinical Study Site, Santa Cecília
  - Clinical Study Site, São José do Rio Preto
  - Clinical Study Site #3, São Paulo
  - Clinical Study Site #4, São Paulo
  - Clinical Study Site 1, São Paulo
  - Clinical Study Site 2, São Paulo
- Bulgaria (2):
  - Clinical Study Site, Dobrich
  - Clinical Study Site, Gabrovo
- Chile (4):
  - Clinical Study Site, Recoleta
  - Clinical Study Site, Santiago
  - Clinical Study Site, Temuco
  - Clincial Study Site, Viña del Mar
- China (10):
  - Clinical Study Site, Lanshan, Shandong
  - Clinical Study Site, Guangdong
  - Clinical Study Site, Harbin
  - Clinical Study Site, Linyi
  - Clinical Study Site 1, Shanghai
  - Clinical Study Site 2, Shanghai
  - Clinical Study Site 1, Tianjin
  - Clinical Study Site 2, Tianjin
  - Clinical Study Site, Xuzhou
  - Clinical Study Site, Zhejiang
- Colombia (3):
  - Clinical Study Site, Barranquilla
  - Clinical Study Site, Bogotá
  - Clinical Study Site, Floridablanca
- Czechia (3):
  - Clinical Study Site, Nový Jičín
  - Clinical Study Site, Pelhřimov
  - Clinical Study Site, Prague
- Georgia (7):
  - Clinical Study Site, Batumi
  - Clinical Study Site #6, Tbilisi
  - Clinical Study Site 1, Tbilisi
  - Clinical Study Site 2, Tbilisi
  - Clinical Study Site 3, Tbilisi
  - Clinical Study Site 4, Tbilisi
  - Clinical Study Site 5, Tbilisi
- Greece (10):
  - Clinical Study Site, Pátrai, Achaia
  - Clinical Study Site, Cholargós, Attica
  - Clinical Study Site 1, Athens
  - Clinical Study Site 2, Athens
  - Clinical Study Site 3, Athens
  - Clinical Study Site, Larissa
  - Clinical Study Site, Pylaia
  - Clinical Study Site 1, Thessaloniki
  - Clinical Study Site 2, Thessaloniki
  - Clinical Study Site 3, Thessaloniki
- Hungary (6):
  - Clinical Study Site, Gyula, Bekes County
  - Clinical Study Site, Tatabánya, Komárom-Esztergom
  - Clinical Study Site, Farkasgyepű, Veszprém megye
  - Clinical Study Site, Budapest
  - Clinical Study Site, Debrecen
  - Clinical Study Site, Zalaegerszeg
- Jordan (2):
  - Clinical Study Site, Amman
  - Clinical Study Site, Irbid
- Lebanon (3):
  - Clinical Study Site, Bsalîm
  - Clinical Study Site, Mazraat ech Choûf
  - Clinical Study Site, Sidon
- Malaysia (6):
  - Clinical Study Site, Kampung Baharu Nilai
  - Clinical Study Site #1, Kuala Lumpur
  - Clinical Study Site #2, Kuala Lumpur
  - Clinical Study Site, Kuching
  - Clinical Study Site, Pulau Pinang
  - Clinical Study Site, Tanjong Bungah
- Mexico (9):
  - Clinical Study Site, Coahuila
  - Clinical Study Site, Cuautitlán
  - Clinical Study Site, Jalisco
  - Clinical Study Site, León
  - Clinical Study Site 1, Monterrey
  - Clinical Study Site 2, Monterrey
  - Clinical Study Site 3, Monterrey
  - Clinical Study Site, Oaxaca City
  - Clinical Study Site, San Luis Potosí City
- Philippines (9):
  - Clinical Study Site, Bacolod City
  - Clinical Study Site, Batangas
  - Clinical Study Site, Cebu
  - Clinical Study Site, City of Taguig
  - Clinical Study Site, Davao City
  - Clinical Study Site 1, Manila
  - Clinical Study Site 2, Manila
  - Clinical Study Site #1, Quezon City
  - Clinical Study Site #2, Quezon City
- Poland (12):
  - Clinical Study Site, Dąbrowa Górnicza
  - Clinical Study Site, Gdynia
  - Clinical Study Site, Krakow
  - Clinical Study Site, Lodz
  - Clinical Study Site, Olsztyn
  - Clinical Study Site, Poznan
  - Clinical Study Site, Prabuty
  - Clinical Study Site, Radom
  - Clinical Study Site, Rzeszów
  - Clinical Study Site, Torun
  - Clinical Study Site, Warsaw
  - Clinical Study Site, Wodzisław Śląski
- Romania (5):
  - Clinical Study Site 1, Craiova
  - Clinical Study Site 2, Craiova
  - Clinical Study Site, Floreşti
  - Clinical Study Site, Ploieşti
  - Clinical Study Site, Timișoara
- Russia (25):
  - Clinical Study Site, Ufa, Republic Bashkortost
  - Clinical Study Site, Pushkin, Sankt-Peterburg
  - Clinical Study Site, Arkhangelsk
  - Clinical Study Site, Belgorod
  - Clinical Study Site, Chelyabinsk
  - Clinical Study Site, Kaluga
  - Clinical Study Site, Kazan'
  - Clinical Study Site, Kemerovo
  - Clinical Study Site, Kislino
  - Clinical Study Site, Kursk
  - Clinical Study Site 1, Moscow
  - Clinical Study Site 2, Moscow
  - Clinical Study Site 3, Moscow
  - Clinical Study Site, Omsk
  - Clinical Study Site, Pyatigorsk
  - Clinical Study Site 1, Saint Petersburg
  - Clinical Study Site 2, Saint Petersburg
  - Clinical Study Site 3, Saint Petersburg
  - Clinical Study Site 4, Saint Petersburg
  - Clinical Study Site, Samara
  - Clinical Study Site, Saransk
  - Clinical Study Site, Sochi
  - Clinical Study Site 1, Tomsk
  - Clinical Study Site 2, Tomsk
  - Clinical Study Site, Yekaterinburg
- Spain (3):
  - Clinical Study Site, Manresa, Barcelona
  - Clinical Study Site, Barcelona
  - Clinical Study Site, Pamplona
- Taiwan (11):
  - Clinical Study Site, Chang-hua
  - Clinical Study Site, Hualien City
  - Clinical Study Site 1, Kaohsiung City
  - Clinical Study Site 2, Kaohsiung City
  - Clinical Study Site 1, New Taipei City
  - Clinical Study Site 2, New Taipei City
  - Clinical Study Site 1, Taichung
  - Clinical Study Site 2, Taichung
  - Clinical Study Site 1, Taipei
  - Clinical Study Site 2, Taipei
  - Clinical Study Site 3, Taipei
- Thailand (10):
  - Clinical Study Site, Hat Yai, Changwat Songkhla
  - Clinical Study Site, Lopburi, Muang
  - Clinical Study Site #1, Bangkok
  - Clinical Study Site #2, Bangkok
  - Clinical Study Site, Chiang Rai
  - Clinical Study Site, Khon Kaen
  - Clinical Study Site, Lampang
  - Clinical Study Site, Phitsanulok
  - Clinical Study Site, Ratchathewi
  - Clinical Study Site, Udon Thani
- Turkey (Türkiye) (16):
  - Clinical Study Site 1, Adana
  - Clinical Study Site 2, Adana
  - Clinical Study Site 1, Ankara
  - Clinical Study Site 2, Ankara
  - Clinical Study Site 3, Ankara
  - Clinical Study Site 4, Ankara
  - Clinical Study Site 5, Ankara
  - Clinical Study Site, Edirne
  - Clinical Study Site 1, Istanbul
  - Clinical Study Site 2, Istanbul
  - Clinical Study Site 3, Istanbul
  - Clinical Study Site 4, Istanbul
  - Clinical Study Site 1, Izmir
  - Clinical Study Site 2, Izmir
  - Clinical Study Site 3, Izmir
  - Clinical Study Site, Samsun
- Ukraine (12):
  - Clinical Study Site, Dnipro
  - Clinical Study Site, Ivano-Frankivsk
  - Clinical Study Site, Kharkiv
  - Clinical Study Site, Kherson
  - Clinical Study Site 1, Kiev
  - Clinical Study Site 2, Kiev
  - Clinical Study Site, Kirovohrad
  - Clinical Study Site 1, Kyiv
  - Clinical Study Site 2, Kyiv
  - Clinical Study Site, Uzhhorod
  - Clinical Study Site, Vinnytsia
  - Clinical Study Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Perez J, Kerr KM, Baker B, Fang F, Li J, McDonald J, Li S, Gao B, Pouliot JF, Seebach F, Lowy I, Gullo G, Herman G, Hamilton J, Rietschel P, McGuire K. Clinical Interchangeability of PD-L1 Immunohistochemistry Assays in First-Line Non-Small Cell Lung Cancer Management With Cemiplimab. JCO Precis Oncol. 2025 Sep;9:e2500177. doi: 10.1200/PO-25-00177. Epub 2025 Sep 24. PMID 40991883
- [Derived] Ozguroglu M, Kilickap S, Sezer A, Gumus M, Bondarenko I, Gogishvili M, Nechaeva M, Schenker M, Cicin I, Ho GF, Kulyaba Y, Zyuhal K, Scheusan RI, Garassino MC, He X, Kaul M, Okoye E, Li Y, Li S, Pouliot JF, Seebach F, Lowy I, Gullo G, Rietschel P. First-line cemiplimab monotherapy and continued cemiplimab beyond progression plus chemotherapy for advanced non-small-cell lung cancer with PD-L1 50% or more (EMPOWER-Lung 1): 35-month follow-up from a mutlicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2023 Sep;24(9):989-1001. doi: 10.1016/S1470-2045(23)00329-7. Epub 2023 Aug 14. PMID 37591293
- [Derived] Gumus M, Chen CI, Ivanescu C, Kilickap S, Bondarenko I, Ozguroglu M, Gogishvili M, Turk HM, Cicin I, Harnett J, Mastey V, Naumann U, Reaney M, Konidaris G, Sasane M, Brady KJS, Li S, Gullo G, Rietschel P, Sezer A. Patient-reported outcomes with cemiplimab monotherapy for first-line treatment of advanced non-small cell lung cancer with PD-L1 of >/=50%: The EMPOWER-Lung 1 study. Cancer. 2023 Jan 1;129(1):118-129. doi: 10.1002/cncr.34477. Epub 2022 Oct 29. PMID 36308296
- [Derived] Sezer A, Kilickap S, Gumus M, Bondarenko I, Ozguroglu M, Gogishvili M, Turk HM, Cicin I, Bentsion D, Gladkov O, Clingan P, Sriuranpong V, Rizvi N, Gao B, Li S, Lee S, McGuire K, Chen CI, Makharadze T, Paydas S, Nechaeva M, Seebach F, Weinreich DM, Yancopoulos GD, Gullo G, Lowy I, Rietschel P. Cemiplimab monotherapy for first-line treatment of advanced non-small-cell lung cancer with PD-L1 of at least 50%: a multicentre, open-label, global, phase 3, randomised, controlled trial. Lancet. 2021 Feb 13;397(10274):592-604. doi: 10.1016/S0140-6736(21)00228-2. PMID 33581821